CLINICAL TRIAL: NCT05531331
Title: The Effect of Education Via Video Conferencing at Home on Self-Efficacy and Adaptation to Stoma of Individuals With Stoma
Brief Title: The Effect of Education on Self-Efficacy and Adaptation to Stoma of Individuals With Stoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Edanur Ozkaya, Student of master's degree, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 56786525-050.04.04/236864
Record Dates: First submitted 2022-09-05; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Stoma Ileostomy; Stoma Colostomy; Self Efficacy; Adjustment; Colorectal Cancer; Colorectal Disorders
Keywords: Adaptation, Colostomy, Education, Ileostomy, Self-Efficacy
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is a parallel group randomized controlled study.
Masking Description: Masking was not performed in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): After discharge, the individuals in the experimental group were given training by the researcher through training booklets prepared by the Association of Wound Ostomy Incontinence Nurses and video conference in four interviews. The first interview was done on the 5th day after discharge, the second on the 10th day, the third on the 15th day, and the fourth on the 2nd month.
  Interventions: Behavioral: At home education via video conferencing
- Control Group (No Intervention): Individuals with stoma in the control group received the training of the company representative that sells stoma materials routinely in the hospital.

INTERVENTIONS:
Behavioral: At home education via video conferencing — Educational booklets are given according to the type of stoma. The individual with the stoma was told that the researcher was always reachable by phone and could communicate if he had any problems. The individuals with stoma in the experimental group received the training of the company representative that sells stoma materials, which is routinely given in the hospital. After discharge, training was given by the researcher via video conference in a total of four interviews. The first interview was done on the 5th day after discharge, the second on the 10th day, the third on the 15th day, and the fourth on the 2nd month. A post-test was conducted at the end of the 4th training interview, which was administered via video conferencing.
  Arms: Intervention Group

SUMMARY:
The aim of this study is to determine the effect of stoma care training given at home via videoconferencing after discharge on the self-efficacy and compliance with stoma of individuals with stoma. In addition to the main purpose, it is aimed to determine whether stoma care education given via video conference at home has an effect on individuals with stoma to perform their own stoma care.

DETAILED DESCRIPTION:
After discharge, the individuals in the experimental group were given training by the researcher through training booklets prepared by the Association of Wound Ostomy Incontinence Nurses and video conference in four interviews. The first interview was done on the 5th day after discharge, the second on the 10th day, the third on the 15th day, and the fourth on the 2nd month. Individuals with stoma in the control group received the training routinely given in the hospital. Self-efficacy and compliance with stoma were measured at baseline and at 2 months. The ability to care for one's own stoma was evaluated at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Opening stoma for the first time,
* Stoma opening surgery Dr. Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital, 3rd Floor Surgical Oncology Clinic,
* Whether the opened stoma is a colostomy or an ileostomy,
* Able to speak and understand Turkish,
* be over 18 years old,
* Not having any mental problems that prevent them from being trained and practiced on stoma care,
* Not having an obstacle to performing stoma care on their own in terms of vision, hearing and motor skills,
* Possibility of meeting via video conference,
* He voluntarily agrees to participate in the research.

Exclusion Criteria:

* Previous stoma opening experience,
* Not being discharged within 10 days after the operation,
* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
The change in the self-efficacy of the experimental group according to the Stoma Self-Efficacy Scale scores at the end of the second month | Baseline, 2nd month
  The Stoma Self-Efficacy Scale was developed to measure self-efficacy in individuals with stoma. The scale was developed by Bekkers et al. (1996). It is a 22-item scale with two sub-dimensions. Items in this scale are in 5-point Likert type. The first sub-dimension is the "Stoma Care Self-Efficacy" sub-dimension, which consists of the first 13 items. The second sub-dimension is the "Social Self-Efficacy" sub-dimension consisting of the remaining nine items. The minimum score that can be taken from the scale is 22, the maximum score is 110, and an increase in the score from the scale indicates high levels of self-efficacy. There is no reverse scored item in the scale.
The change in the adaptation of the experimental group according to the Ostomy Adjustment Inventory-23 scores at the end of the second month | Baseline, 2nd month
  It was created by Maekawa (2000) and later this scale was arranged by Simmons et al. (2009) in the form of Ostomy Adjustment Scale-23, consisting of 23 items and 4 sub-dimensions. OAS-23, a self-assessment scale, is a scale used to evaluate the level of adjustment in individuals with stoma. 4 sub-dimensions in this scale: accepting (includes items 1, 3, 4, 6, 9, 14, 15, 19, 23.), anxiety/worry (12, 13, 17, 20, 21 items) .), social cohesion (includes items 5, 7, 8, 11), and anger (includes items 2 and 10). At the same time, there are 3 items (16, 18 and 22) that are not included in any sub-dimensions. Each item of the scale is evaluated in a 5-point Likert type.

SECONDARY OUTCOMES:
The change in the ability of individuals with stoma to care for their stoma at the end of the 2nd month | Baseline, 2nd month
  After the individuals with stoma in the experimental group were trained by the researcher throughout the study, it was evaluated that they could or could not perform their own stoma care under the supervision of the researcher. However, the status of individuals in the control group for maintaining stoma care is based on their own statements.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz HARPUTLU, PhD, RN, Study Director — Ankara University
Locations (1):
- Edanur Özkaya, Pamukkale, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will share.
Supporting Information: Study Protocol, SAP
Time Frame: starting 1 months after publication
Access Criteria: all people access

REFERENCES:
- [Result] Dinuzzi VP, Palomba G, Minischetti M, Amendola A, Aprea P, Luglio G, De Palma GD, Aprea G. Telemedicine in Patients With an Ostomy During the COVID-19 Pandemic: A Retrospective Observational Study. Wound Manag Prev. 2021 Jan;67(1):12-17. PMID 33448938
- [Result] Jin Y, Ma H, Jimenez-Herrera M. Self-disgust and stigma both mediate the relationship between stoma acceptance and stoma care self-efficacy. J Adv Nurs. 2020 Oct;76(10):2547-2558. doi: 10.1111/jan.14457. Epub 2020 Jul 23. PMID 32700799
- [Result] Krogsgaard M, Kristensen HO, Furnee EJB, Verkuijl SJ, Rama NJ, Domingos H, Maciel J, Solis-Pena A, Espin-Basany E, Hidalgo-Pujol M, Biondo S, Sjovall A, Emmertsen KJ, Thyo A, Christensen P. Life with a stoma across five European countries-a cross-sectional study on long-term rectal cancer survivors. Support Care Cancer. 2022 Nov;30(11):8969-8979. doi: 10.1007/s00520-022-07293-y. Epub 2022 Aug 5. PMID 35930059
- [Result] Nam KH, Kim HY, Kim JH, Kang KN, Na SY, Han BH. Effects of social support and self-efficacy on the psychosocial adjustment of Korean ostomy patients. Int Wound J. 2019 Mar;16 Suppl 1(Suppl 1):13-20. doi: 10.1111/iwj.13038. PMID 30793862
- [Result] Seo HW. Effects of the frequency of ostomy management reinforcement education on self-care knowledge, self-efficacy, and ability of stoma appliance change among Korean hospitalised ostomates. Int Wound J. 2019 Mar;16 Suppl 1(Suppl 1):21-28. doi: 10.1111/iwj.13047. PMID 30793857
- [Result] Wang QQ, Zhao J, Huo XR, Wu L, Yang LF, Li JY, Wang J. Effects of a home care mobile app on the outcomes of discharged patients with a stoma: A randomised controlled trial. J Clin Nurs. 2018 Oct;27(19-20):3592-3602. doi: 10.1111/jocn.14515. Epub 2018 Jul 10. PMID 29775491
- [Result] Wen SL, Li J, Wang AN, Lv MM, Li HY, Lu YF, Zhang JP. Effects of transtheoretical model-based intervention on the self-management of patients with an ostomy: A randomised controlled trial. J Clin Nurs. 2019 May;28(9-10):1936-1951. doi: 10.1111/jocn.14731. Epub 2019 Feb 18. PMID 30549366
- [Result] White T, Watts P, Morris M, Moss J. Virtual Postoperative Visits for New Ostomates. Comput Inform Nurs. 2019 Feb;37(2):73-79. doi: 10.1097/CIN.0000000000000498. PMID 30562169
- [Result] Yan MH, Lv L, Zheng MC, Jin Y, Zhang JE. Quality of Life and Its Influencing Factors Among Chinese Patients With Permanent Colostomy in the Early Postoperative Stage: A Longitudinal Study. Cancer Nurs. 2022 Jan-Feb 01;45(1):E153-E161. doi: 10.1097/NCC.0000000000000893. PMID 33003121
- [Result] Zhang JE, Wong FK, You LM, Zheng MC, Li Q, Zhang BY, Huang MR, Ye XM, Liang MJ, Liu JL. Effects of enterostomal nurse telephone follow-up on postoperative adjustment of discharged colostomy patients. Cancer Nurs. 2013 Nov-Dec;36(6):419-28. doi: 10.1097/NCC.0b013e31826fc8eb. PMID 23051876
- [Derived] Ozkaya E, Harputlu D. The Effect of Education Via Videoconferencing at Home on Individuals' Self-efficacy and Adaptation to Life with a Stoma: A Randomized Controlled Study. Adv Skin Wound Care. 2024 Feb 1;37(2):86-94. doi: 10.1097/ASW.0000000000000098. PMID 38241451